CLINICAL TRIAL: NCT01974427
Title: Functional Brain Imaging in Healthy Volunteers to Study Cognitive Functions
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140002; 14-N-0002
Record Dates: First submitted 2013-10-26; First posted 2013-11-01 (Estimated); Last update posted 2019-05-31 (Actual); Status verified 2019-05-29

CONDITIONS: Healthy Volunteers
Keywords: Magnetic Resonance Imaging (MRI); Functional Imaging; BOLD Effect; EEG; MEG

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Objective:

The goal of this protocol is to improve understanding scale-free brain activity and conscious vs. unconscious processing by performing small behavioral, electrophysiological, neuroimaging and brain stimulation pilot substudies. This research is expected to help develop techniques and hypotheses for future research on these topics.

We will conduct:

* Pilot Substudy: Pilot substudies are exploratory in nature, in order to develop enough information to generate a hypothesis. The criterion for transition to a new full protocol will be acquisition of sufficient information to generate a power analysis. There are no enrollment limitations for pilot substudies.
* Hypothesis-Testing Substudy is defined as a study with a specific hypothesis to be tested that can be completed with a few healthy volunteers or patients. Hypothesis-testing substudies will undergo statistical and PIRC reviews after 6 subjects (if there is one group) or after 12 (6 per arm) if two groups are studied before additional subjects are recruited. In the event of subject dropout or unsuccessful recording, replacement will be recruited. Together, the P.I. and PIRC will decide whether to continue the hypothesis substudy with more subjects without an amendment or whether an amendment or new protocol would be necessary. A memo requesting a review of hypothesis-testing substudies for possible additional enrollment will be sent to PIRC and the statistical reviewer. The memo will be forwarded to the CNS IRB.
* Technical development of new experimental paradigms and data analysis methods.

This protocol includes only non-invasive techniques with minimal risk (MRI, EEG, MEG, EMG, tDCS).

Study Population:

We plan to recruit up to 120 healthy volunteers aged 18-65.

Design:

We will design small projects that are pertinent to the theme of scale-free brain activity and conscious/unconscious processing. We will investigate healthy volunteers in the resting state or while they perform simple motor or sensory tasks. If a hypothesis testing substudy leads to results of interest and if a larger population is necessary to reach statistical significance, a separate protocol will be submitted with a priori hypotheses, specific study design and power analysis adapted from the pilot or exploratory substudies performed in the present protocol.

In the substudies, brain activity of healthy human volunteers will be monitored by functional magnetic resonance imaging (fMRI), magnetoencephalography (MEG), electroencephalography (EEG), or simultaneous MEG-EEG. Anatomical MRI will be collected in some subjects to allow better localization of brain dynamics. Because transcranial direct-current stimulation (tDCS) is ideally suited to modulate the slow component of scale-free brain activity, we will also investigate the effect of tDCS on brain activity and/or behavioral performance in cognitive tasks. tDCS will be administered sequentially, but not simultaneously, with brain-activity monitoring by fMRI/MEG/EEG. Most experiments will be conducted in conjunction with cognitive tasks. In some experiments, we will study resting-state brain function, during which spontaneous brain activity is collected without a specific externally administered task.

Outcome Measures:

MRI: to analyze measures such as the anatomical structures of the brain (using structural MRI); amplitude of the blood-oxygenation-level-dependent (BOLD) signal (using fMRI); cerebral blood flow [using arterial spin labeling (ASL)] and different neurotransmitter levels in brain regions of interest [using magnetic resonance spectroscopy (MRS)].

EEG and MEG: to quantify measures such as power spectrum, event- or task-related potentials, synchronization/desynchronization, and coherence between sensors or sources located close to the brain areas of interest.

tDCS: to analyze changes in behavioral measures and/or fMRI/EEG/MEG activity caused by tDCS.

Behavioral measures: to quantify measures such as hit rate, reaction times, electromyography (EMG) patterns.

We may measure autonomic data during the course of the experiment (such as heart rate, respiration, end-tidal CO2, skin conductance), which will be correlated with the outcome measures.

DETAILED DESCRIPTION:
Objective:

The goal of this protocol is to improve understanding scale-free brain activity and conscious vs. unconscious processing by performing small behavioral, electrophysiological, neuroimaging and brain stimulation pilot substudies. This research is expected to help develop techniques and hypotheses for future research on these topics.

We will conduct:

* Pilot Substudy: Pilot substudies are exploratory in nature, in order to develop enough information to generate a hypothesis. The criterion for transition to a new full protocol will be acquisition of sufficient information to generate a power analysis. There are no enrollment limitations for pilot substudies.
* Hypothesis-Testing Substudy is defined as a study with a specific hypothesis to be tested that can be completed with a few healthy volunteers or patients. Hypothesis-testing substudies will undergo statistical and PIRC reviews after 6 subjects (if there is one group) or after 12 (6 per arm) if two groups are studied before additional subjects are recruited. In the event of subject dropout or unsuccessful recording, replacement will be recruited. Together, the P.I. and PIRC will decide whether to continue the hypothesis substudy with more subjects without an amendment or whether an amendment or new protocol would be necessary. A memo requesting a review of hypothesis-testing substudies for possible additional enrollment will be sent to PIRC and the statistical reviewer. The memo will be forwarded to the CNS IRB.
* Technical development of new experimental paradigms and data analysis methods.

This protocol includes only non-invasive techniques with minimal risk (MRI, EEG, MEG, EMG, tDCS).

Study Population:

We plan to recruit up to 200 healthy volunteers aged 18-65.

Design:

We will design small projects that are pertinent to the theme of scale-free brain activity and conscious/unconscious processing. We will investigate healthy volunteers in the resting state or while they perform simple motor or sensory tasks. If a hypothesis testing substudy leads to results of interest and if a larger population is necessary to reach statistical significance, a separate protocol will be submitted with a priori hypotheses, specific study design and power analysis adapted from the pilot or exploratory substudies performed in the present protocol.

In the substudies, brain activity of healthy human volunteers will be monitored by functional magnetic resonance imaging (fMRI), magnetoencephalography (MEG), electroencephalography (EEG), or simultaneous MEG-EEG. Anatomical MRI will be collected in some subjects to allow better localization of brain dynamics. Because transcranial direct-current stimulation (tDCS) is ideally suited to modulate the slow component of scale-free brain activity, we will also investigate the effect of tDCS on brain activity and/or behavioral performance in cognitive tasks. tDCS will be administered sequentially, but not simultaneously, with brain-activity monitoring by fMRI/MEG/EEG. Most experiments will be conducted in conjunction with cognitive tasks. In some experiments, we will study resting-state brain function, during which spontaneous brain activity is collected without a specific externally administered task.

Outcome Measures:

MRI: to analyze measures such as the anatomical structures of the brain (using structural MRI); amplitude of the blood-oxygenation-level-dependent (BOLD) signal (using fMRI); cerebral blood flow [using arterial spin labeling (ASL)] and different neurotransmitter levels in brain regions of interest [using magnetic resonance spectroscopy (MRS)].

EEG and MEG: to quantify measures such as power spectrum, event- or task-related potentials, synchronization/desynchronization, and coherence between sensors or sources located close to the brain areas of interest.

tDCS: to analyze changes in behavioral measures and/or fMRI/EEG/MEG activity caused by tDCS.

Behavioral measures: to quantify measures such as hit rate, reaction times, electromyography (EMG) patterns.

We may measure autonomic data during the course of the experiment (such as heart rate, respiration, end-tidal CO2, skin conductance), which will be correlated with the outcome measures.

ELIGIBILITY:
* INCLUSION CRITERIA:

A subject can be included if he/she:

is in good general health;

is between 18 and 65 years old;

is capable of understanding the procedures and requirements of this study;

is willing and able to provide his/her own informed consent.

EXCLUSION CRITERIA:

A subject will be excluded if he/she:

has a contraindication to MR scanning such as the following: pregnancy, aneurysm clip; implanted neural stimulator; implanted cardiac pacemaker or auto-defibrillator; cochlear implant; ocular foreign body (e.g. metal shavings); insulin pump as per the NMR Safety Screening Form.

underwent brain surgery, who have a central nervous system illness, neurological lesion, a psychiatric history or recurrent migraines that require medication will also be excluded from this study: Healthy volunteer form.

has uncontrolled medical problems, such as diabetes mellitus, hypertension, pulmonary or airway disease, heart failure, coronary artery disease.

has metal in the cranial cavity and/or holes in the skull made by trauma or surgery.

cannot lie comfortably flat on their back for up to 180 minutes in the MRI scanner

has claustrophobia

Subjects may participate in this study, but will not be allowed to have a 7T MRI scan if they have metallic dental crowns or a bridge.

Subjects may participate in the study, but will not have tDCS if they have broken skin or a wound in the area where electrodes will be placed.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2013-10-26; Primary Completion 2018-06-20 (Actual); Study Completion 2018-06-20 (Actual)

PRIMARY OUTCOMES:
Behavioral measures, brain activity recorded by MRI, EEG, MEG, as well as changes in the above measures induced by tDCS | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Alan P. Koretsky, Ph.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] He BJ, Zempel JM, Snyder AZ, Raichle ME. The temporal structures and functional significance of scale-free brain activity. Neuron. 2010 May 13;66(3):353-69. doi: 10.1016/j.neuron.2010.04.020. PMID 20471349
- [Background] He BJ. Scale-free properties of the functional magnetic resonance imaging signal during rest and task. J Neurosci. 2011 Sep 28;31(39):13786-95. doi: 10.1523/JNEUROSCI.2111-11.2011. PMID 21957241
- [Background] Ray S, Maunsell JH. Different origins of gamma rhythm and high-gamma activity in macaque visual cortex. PLoS Biol. 2011 Apr;9(4):e1000610. doi: 10.1371/journal.pbio.1000610. Epub 2011 Apr 12. PMID 21532743